CLINICAL TRIAL: NCT04313101
Title: Association Between Thyroid Dysfunction and Intensive Care Unit Acquired Weakness: A Case Control Study
Brief Title: Association Between Thyroid Dysfunction and Intensive Care Unit Acquired Weaknesss
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tarek Samir Shabana, Tarek Samir Shabana, Ain Shams University
Other Study IDs: FMASU R 10/2020
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Thyroid Abnormalities; ICU Acquired Weakness
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cases (ICUAW): 57 critically ill patients developing ICUAW during their stay in the intensive care unit will be included in the study as cases.
  Interventions: Other: withdrawl of blood samples for thyroid function testing
- Controls: A total of 57 Critically ill patients in the same period who did not develop ICU acquired weakness during their ICU stay will be included as controls.
  Interventions: Other: withdrawl of blood samples for thyroid function testing

INTERVENTIONS:
Other: withdrawl of blood samples for thyroid function testing — Blood samples will be withdrawn from patients admitted to the intensive care for more than 7 days to measure Thyroid hormones (Free T3: Tri-iodothyronine and Free T4:thyroxine) and TSH ( Thyroid Stimulating Hormone) using ELISA kits. Reference ranges will be as follows: TSH 0.4-4mU/L, Free T3 2-4.4 mU/L, Free T4 0.8-1.9 mU/L. Patients will be then categorized into one of the following categories
  * Euthyroid ( Normal TSH, FT3 and FT4)
  * Hyperthyroid (Low TSH) either overt (increased FT3 and /or FT4) or subclinical (normal FT4 and FT3).
  * Hypothyroid (Elevated TSH) either overt (Low FT3 and FT4) or subclinical (Normal FT3 and FT4)
  * Non-thyroidal illness syndrome : normal or low TSH in addition to low FT3 ± Low FT4 levels.

SUMMARY:
Intensive care unit-acquired weakness (ICU-AW) is the most common neuromuscular impairment in critically ill patients. It affects more than 50 % of patients in the intensive care and is related to many problems as difficult weaning from mechanical ventilation, prolonged hospital stay and increased mortality.Thyroid disorders are also associated with neuromuscular abnormalities and may decrease the threshold for the development of any type of myopathy. However, no previous study investigated the direct relationship between thyroid dysfunction and ICUAW.This study aims at evaluation of the association between thyroid dysfunction and intensive care unit acquired weakness.

DETAILED DESCRIPTION:
Intensive care unit acquired weakness refers to muscle weakness encountered in the intensive care unit as a consequence of critical illness. It affects more than 50 % of patients in the intensive care and is related to many problems as difficult weaning from mechanical ventilation, prolonged hospital stay and increased mortality.

There are three distinct entities for ICUAW that can only be differentiated by neurophysiological studies. These are critical illness myopathy (CIM), critical illness polyneuropathy (CIP) and critical illness neuromyopathy (CINM).

Identification of risk factors responsible for the development of ICUAW is the first step in the prevention and management of this disorder. Till time septic shock, hyperglycemia, high dose steroid therapy, prolonged mechanical ventilation and the use of neuromuscular blocking agents are the main accused.

Thyroid disorders are also associated with neuromuscular abnormalities. Unfortunately, the prevalence of thyroid dysfunction in the intensive care is high reaching 90%. Moreover, patients with severe critical illness, who are typically prone to the development of ICUAW, show changes in their thyroid biochemistry namely low T3 levels (with or without low T4 levels) in the presence of normal TSH levels. These changes are collectively known as Non-Thyroidal illness syndrome (previously low T3 syndrome and Euthyroid sick syndrome) which is the most common form of thyroid dysfunction in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes admitted to the general ICU of Ain Shams University Hospitals with critical illness for more than 7 days * Diagnosis of ICU acquired weakness will be made based on clinical criteria for ICUAW and confirmed by nerve conduction studies.

Exclusion Criteria:

* Patients with cerebrovascular accidents, neuromuscular disorders, spine abnormalities, spinal cord or head injuries, CNS tumors, secondary thyroid disorders and electrolyte disturbances were excluded from the study. Patients receiving thyroid replacement or anti-thyroid drugs for the treatment of any throid disorder will be also excluded from the study as these drugs may alter their thyroid biochemistry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical criteria for Intensive care unit acquired weakness :
  1. . Weakness developing after the onset of critical illness
  2. . Generalized (Proximal and distal), symmetrical and flaccid weakness with sparing of cranial nerves
  3. . MRC) score< 48 (or mean score <4 in all tested muscles on more than two occasions more than 24 hours apart) .
  4. . Mechanical ventilator dependence
  5. . Cause of weakness not related directly to the underlying critical illness
     * Final Diagnosis of ICUAW :
       1. Presence of criteria (1), (2) and (5) + (3) Or (4)
       2. Results of Nerve conduction studies
  Nerve conduction studies :Unilateral bedside nerve conduction tests of the sural and peroneal nerves (reduced CMAP amplitudes).
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Association between thyroid dysfunction and ICUAW | Patients admitted to the intensive care for more than 7 days
  Comparison between both groups as regards thyroid functions and the incidence of each of the four categories of thyroid function.Logistic regression will be done to assess each of the four categories of thyroid function as a risk factor in the development of ICUAW in the presence of other risk factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided